CLINICAL TRIAL: NCT02394288
Title: Perioperative High-sensitivity Cardiac Troponin Levels in Healthy Adults Undergoing Elective Trauma Surgery
Brief Title: Perioperative Cardiac Troponin Levels in Healthy Adults
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Andreas Duma, MD, MSc, Medical University of Vienna
Other Study IDs: 1579/2014
Record Dates: First submitted 2015-03-13; First posted 2015-03-20 (Estimated); Last update posted 2016-03-21 (Estimated); Status verified 2016-03

CONDITIONS: Extremity Orthopedic Surgery
Keywords: Cardiac Troponin; Perioperative Period; surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Adults without cardiac disease: Extremity orthopedic or trauma surgery
  Interventions: Procedure: Extremity orthopedic or trauma surgery

INTERVENTIONS:
Procedure: Extremity orthopedic or trauma surgery — hip, leg, shoulder, arm

SUMMARY:
This study will determine the extent of high-sensitivity cardiac troponin (hs-cTn) release in patients without cardiac risk factors undergoing extremity orthopedic surgery. This study will provide important evidence on how to interpret postoperative cardiac troponin elevations.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-35 years
* Extremity orthopedic or trauma surgery: leg, hip, arm, shoulder.
* Planned overnight hospital admission
* No cardiac risk factors (Lee's Revised Cardiac Risk Index Class 1)
* American Society of Anesthesiologists (ASA) physical status I-II

Exclusion Criteria:

* Any history or symptoms of cardiac disease
* Kidney or liver disease
* Recent or current trauma to the trunk or head
* Persons with increased vulnerability (e.g. cognitive limitations, prisoners,…)
* Pregnancy

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients undergoing extremity surgery without history of cardiovascular disease
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2015-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Perioperative change of high-sensitivity cardiac troponin plasma level | 24 hours preoperatively to postoperative day (POD) 1
  3 samples:
  1. Preoperative,
  2. POD 0, and
  3. POD 1

SECONDARY OUTCOMES:
Peak high-sensitivity cardiac troponin plasma level | 24 hours preoperatively to POD 1
  3 samples:
  1. Preoperative,
  2. POD 0, and
  3. POD 1
Incidence rate of high-sensitivity cardiac troponin plasma level elevation | 24 hours preoperatively to POD 1
  3 samples:
  1. Preoperative,
  2. POD 0, and
  3. POD 1

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Duma, MD, MSc, Principal Investigator — Medical University of Vienna
Locations (1):
- Division of General Anaesthesia and Intensive Care Medicine, Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Derived] Duma A, Wagner C, Titz M, Maleczek M, Hupfl M, Weihs VB, Samaha E, Herkner H, Szekeres T, Mittlboeck M, Scott MG, Jaffe AS, Nagele P. High-sensitivity cardiac troponin T in young, healthy adults undergoing non-cardiac surgery. Br J Anaesth. 2018 Feb;120(2):291-298. doi: 10.1016/j.bja.2017.09.001. Epub 2017 Dec 5. PMID 29406178